CLINICAL TRIAL: NCT04165031
Title: A Phase 1/2 Study of LY3499446 Administered to Patients With Advanced Solid Tumors With KRAS G12C Mutation
Brief Title: A Study of LY3499446 in Participants With Advanced Solid Tumors With KRAS G12C Mutation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to an unexpected toxicity finding.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17501; J2K-MC-JZKA (Other: Eli Lilly and Company); 2019-003070-53 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumor; Non-Small Cell Lung Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — abemaciclib; Cetuximab; Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3499446 Phase 1 Cohort A1 High Dose (Experimental): Participants received high dose LY3499446 as oral monotherapy twice daily (BID) in 21-day cycles.
  Interventions: Drug: LY3499446
- LY3499446 Phase 1 Cohort AO Mid Dose (Experimental): Participant received mid dose LY3499446 as oral monotherapy once every other day (QOD) in 21-day cycles.
  Interventions: Drug: LY3499446
- LY3499446 Phase 1 Cohort A-2 Low Dose (Experimental): Participants received low dose LY3499446 as oral monotherapy once daily (QD) in 21-Day cycles.
  Interventions: Drug: LY3499446
- LY3499446 + Combination Drugs Phase 1 (Experimental): LY3499446 combined with either abemaciclib (orally), erlotinib (orally), or cetuximab (IV).
  This trial was terminated prior to initiation of combination therapy cohorts.
  Interventions: Drug: LY3499446; Drug: Abemaciclib; Drug: Cetuximab; Drug: Erlotinib
- LY3499446 Monotherapy + Combination Drugs Phase 2 (Experimental): LY3499446 as oral monotherapy and LY3499446 combined with either abemaciclib (orally), erlotinib (orally), or cetuximab (IV).
  The trial was terminated prior to initiation of Phase 2 of this study.
  Interventions: Drug: LY3499446; Drug: Abemaciclib; Drug: Cetuximab; Drug: Erlotinib
- Docetaxel Phase 2 (Active Comparator): Docetaxel IV infusion.
  The trial was terminated prior to initiation of Phase 2 of this study.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: LY3499446 — Administered orally
  Arms: LY3499446 + Combination Drugs Phase 1; LY3499446 Monotherapy + Combination Drugs Phase 2; LY3499446 Phase 1 Cohort A-2 Low Dose; LY3499446 Phase 1 Cohort A1 High Dose; LY3499446 Phase 1 Cohort AO Mid Dose
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: LY3499446 + Combination Drugs Phase 1; LY3499446 Monotherapy + Combination Drugs Phase 2
Drug: Cetuximab — Administered IV
  Arms: LY3499446 + Combination Drugs Phase 1; LY3499446 Monotherapy + Combination Drugs Phase 2
Drug: Erlotinib — Administered orally
  Arms: LY3499446 + Combination Drugs Phase 1; LY3499446 Monotherapy + Combination Drugs Phase 2
Drug: Docetaxel — Administered IV
  Arms: Docetaxel Phase 2

SUMMARY:
The reason for this study is to see if the study drug LY3499446 is safe and effective in participants with solid tumors with KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have diagnosis of a solid tumor with KRAS G12C mutation that did not respond to at least 1 line of standard therapy and has spread to other part(s) of the body
* For phase II, participants must be willing to have new tumor tissue biopsies (doctor removes a small amount of tissue) during the study if it does not cause undue risks to health
* Participants must be willing to use highly effective birth control
* Participants must have adequate organ function
* Participants must be able to swallow capsules

Exclusion Criteria:

* Participants must not have certain infections such as hepatitis or tuberculosis or HIV that is not well controlled
* Participants must not have another serious medical condition including a serious heart condition, such as congestive heart failure, unstable angina pectoris, or heart attack within the last three months
* Participants must not have cancer of the central nervous system that is not stable
* Participants must not be pregnant or breastfeeding
* Participants must not use herbal supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (4):
  - Indiana Univ Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (2):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Linear Clinical Research Ltd, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3499446 in Participants With Advanced Solid Tumors With KRAS G12C Mutation — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JZKA#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was identified as having completed the study if the participant was observed until event of progressive disease (PD) or death, or the participant had discontinued study treatment and is in follow up at the time of the final analysis.
  The study was terminated due to an unexpected toxicity finding.
Groups:
- LY3499446 Phase 1 Cohort A1 (High Dose): Participants received high dose LY3499446 as oral monotherapy twice daily (BID) in 21-day cycles.
- LY3499446 Phase 1 Cohort AO (Mid Dose): Participant received mid dose LY3499446 as oral monotherapy once every other day (QOD) in 21-day cycles.
- LY3499446 Phase 1 Cohort A-2 (Low Dose): Participants received low dose LY 3499446 as oral monotherapy once daily (QD) in 21-day cycles.
- LY3499446 + Combination Drug Phase 1: LY3499446 combined with either abemaciclib (orally), erlotinib (orally), or cetuximab (IV).
  The trial was terminated prior to initiation of this portion.
- LY3499446 Monotherapy + Combination Drug Phase 2: LY3499446 monotherapy orally. LY3499446 combined with either abemaciclib (orally), erlotinib (orally), or cetuximab (IV).
  The trial was terminated prior to initiation of this portion.
- Docetaxel Phase 2: Docetaxel IV infusion.
  The trial was terminated prior to initiation of this portion.
Period: Overall Study
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose) | LY3499446 + Combination Drug Phase 1 | LY3499446 Monotherapy + Combination Drug Phase 2 | Docetaxel Phase 2
Started | 2 | 1 | 2 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 2 | 1 | 2 | 0 | 0 | 0
Completed | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug
Groups:
- LY3499446 Phase 1 Cohort A1 (High Dose): Participants received high dose LY3499446 as oral monotherapy BID in 21-day cycles.
- LY3499446 Phase 1 Cohort AO (Mid Dose): Participant received mid dose LY3499446 as oral monotherapy once QOD in 21-day cycles.
- LY3499446 Phase 1 Cohort A-2 (Low Dose): Participants received low dose LY 3499446 as oral monotherapy once QD in 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose) | LY3499446 + Combination Drug Phase 1 | LY3499446 Monotherapy + Combination Drug Phase 2 | Docetaxel Phase 2 | Total
Number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 0 | 0 | 1
  >=65 years | 1 | 1 | 2 | 0 | 0 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 0 | 0 | 0 | 4
  Male | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 0 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 2 | 0 | 0 | 0 | 5
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Australia | 2 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number or Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is defined as an event that is clinically significant and not clearly related to disease progression or intercurrent illness that occurred within the DLT observation period of the Cycle 1 timeframe.
Time Frame: Cycle 1 (21 Day Cycle)
Population: All participants who received at least one dose of study drug and had a dose limiting toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- LY3499446 Phase 1 Cohort A-2 (Low Dose): Participants received low dose LY3499446 as oral monotherapy once QD in 21-day cycles.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 2 | 1 | 2
Participants | 2 | 1 | 1

2. Primary Outcome: Phase 2: Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR) in Colorectal Cancer (CRC) Cohorts and Other Tumors Cohort
Description: ORR is defined as percentage of participants who achieved a CR or PR out of all the participants treated. Tumor responses were measured and record using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST) v1.1 guidelines. CR is defined as the disappearance of all targeted and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions and no appearance of new lesions.
Time Frame: Baseline through Measured Progressive Disease
Population: Zero participants were analyzed due to early termination of study.
Groups:
- LY3499446 Monotherapy + Combination Drugs Phase 2: LY3499446 combined with either abemaciclib (orally), erlotinib (orally), or cetuximab (IV).
- Docetaxel Phase 2: Docetaxel IV infusion.
Arm/Group | LY3499446 Monotherapy + Combination Drugs Phase 2 | Docetaxel Phase 2
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Phase 2: Progression-Free Survival (PFS) Non-Small Lung Cancer (NSCLC Cohorts)
Description: PFS was defined as the time from study enrollment (for non-randomized cohorts)/ the time from randomization (for randomized cohorts) to the first observation of progressive disease (PD) or death without documented disease progression per RECIST V1.1 criteria.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause
Population: Zero participants were analyzed due to early termination of study.
Arm/Group | LY3499446 Monotherapy + Combination Drugs Phase 2 | Docetaxel Phase 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1: Pharmacokinetics (PK): Average Concentration of LY3499446
Description: Average concentration after the first dose of LY3499446.
Time Frame: Cycle 1 Day 1: Predose, 0.5, 1, 1.5, 2, 3, 4, 8, 24 hours post-dose
Population: All participants who have received at least one dose of study drug and had evaluable PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 2 | 1 | 2
nanograms per milliliter (ng/mL) | NA (NA) — N=2: Geometric mean and Geometric Coefficient of Variation were not calculated, individual values reported:1056 ng/mL and 570 ng/mL. | NA (NA) — N=1: Geometric mean and Geometric Coefficient of Variation were not calculated, individual values reported: 865 ng/mL. | NA (NA) — N=2: Geometric mean and Geometric Coefficient of Variation were not calculated, individual values reported: 225 ng/mL and 116 ng/mL.

5. Secondary Outcome: Phase 1: PK: Average Concentration at Steady State of LY3499446 in Combination With Abemaciclib
Description: PK: Average Concentration at Steady State of LY3499446 in Combination with Abemaciclib
Time Frame: Predose Cycle 1 Day 1 through Cycle 3 Day 1 (21 Day Cycles)
Population: Zero participants were analyzed due to early termination of study.
Groups:
- LY3499446 and Abemaciclib Phase 1: LY3499446 in combination with abemaciclib orally.
Arm/Group | LY3499446 and Abemaciclib Phase 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1: PK: Average Concentration at Steady State of LY3499446 in Combination With Cetuximab
Description: PK: Average Concentration at Steady State of LY3499446 in Combination with Cetuximab
Time Frame: Predose Cycle 1 Day 1 through Cycle 3 Day 1 (21 Day Cycles)
Population: Zero participants were analyzed due to early termination of study.
Groups:
- LY3499446 and Cetuximab Phase 1: LY3499446 in combination with cetuximab intravenously (IV).
Arm/Group | LY3499446 and Cetuximab Phase 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1: PK: Average Concentration at Steady State of LY3499446 in Combination With Erlotinib
Description: PK: Average Concentration at Steady State of LY3499446 in Combination with Erlotinib
Time Frame: Predose Cycle 1 Day 1 through Cycle 3 Day 1 (21 Day Cycles)
Population: Zero participants were analyzed due to early termination of study.
Groups:
- LY3499446 Monotherapy and Erlotinib Phase 1: LY3499446 in combination with erlotinib orally.
Arm/Group | LY3499446 Monotherapy and Erlotinib Phase 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 1: ORR: Percentage of Participants Who Achieve CR or PR
Description: as for outcome 2
Time Frame: Baseline through Measured Progressive Disease (Up to 11 Months)
Population: Zero participants were analyzed due to early termination of study.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Phase 1: PFS
Description: PFS was defined as the time from study enrollment (for non-randomized cohorts)/ the time from randomization (for randomized cohorts) to the first observation of progressive disease (PD) overall response or death without documented disease progression per RECIST V1.1 criteria.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Up to 11 Months)
Population: Zero participants were analyzed due to early termination of study.
Groups:
- LY3499446 Phase 1 Cohort AO (Mid Dose): Participant received mid dose LY3499446 as oral monotherapy QOD in 21-day cycles.
- LY3499446 Phase 1 Cohort A-2 (Low Dose): Participants received low dose LY3499446 as oral monotherapy QD in 21-day cycles in 21-day cycles.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Phase 1: Duration of Response (DoR)
Description: DoR was defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST v1.1 criteria, or the date of death from any cause in the absence of objectively determined disease progression or recurrence.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Up to 11 Months)
Population: Zero participants were analyzed due to early termination of study.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Phase 1: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and SD
Description: DCR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed CR, confirmed PR, or SD out of all participants treatment. Best response is determined from a sequence of responses assessed. Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR. CR is defined as the disappearance of all targeted and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions and no appearance of new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up to 11 Months)
Population: Zero participants were analyzed due to early termination of study.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 11 months
Description: All participants who received at least one dose of study drug.
Groups:
- LY3499446 Phase 1 Cohort A-2 (Low Dose): Participants received low dose LY3499446 as monotherapy orally once QD in 21-day cycles.
Arm/Group | LY3499446 Phase 1 Cohort A1 (High Dose) | LY3499446 Phase 1 Cohort AO (Mid Dose) | LY3499446 Phase 1 Cohort A-2 (Low Dose)
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3499446 Phase 1 Cohort A1 (High Dose) (N=2) | LY3499446 Phase 1 Cohort AO (Mid Dose) (N=1) | LY3499446 Phase 1 Cohort A-2 (Low Dose) (N=2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3499446 Phase 1 Cohort A1 (High Dose) (N=2) | LY3499446 Phase 1 Cohort AO (Mid Dose) (N=1) | LY3499446 Phase 1 Cohort A-2 (Low Dose) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to an unexpected toxicity finding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04165031/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT04165031/SAP_001.pdf